CLINICAL TRIAL: NCT04615754
Title: Ketone Administration in Patients With Pulmonary Hypertension - Effects on Hemodynamics
Brief Title: Ketones for Pulmonary Hypertension - Effects on Hemodynamics
Acronym: KEPAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1-10-72-232-19
Record Dates: First submitted 2020-08-10; First posted 2020-11-04 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Hypertension; Ketonemia
Keywords: Right sided heart catheterization; Echocardiography; Hemodynamics
MeSH Terms: conditions — Hypertension, Pulmonary; Ketosis

STUDY DESIGN:
Intervention Model Description: Randomized cross-over I.e. Ketone infusion is compared to saline infusion in a randomised cross-ove design.
  (Ketones are considered dietary supplement as glucose or lipids)
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and the endpoint-assessor will be masked to intevention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-OHB vs Saline (Experimental): 3-OHB will be infused for 2.5 hours in IPAH (n=5) and CETPH (n=5) patients- 6 in each group is recruited for taking drop-out into account
  Interventions: Dietary Supplement: Hyperketonemia - use of ketone (3-OHB) infusion; Dietary Supplement: Placebo - use of saline infusion
- Saline vs 3-OHB (Experimental): Saline will be infused for 2.5 hours in IPAH (n=5) and CETPH (n=5) patients- 6 in each group is recruited for taking drop-out into account
  Interventions: Dietary Supplement: Hyperketonemia - use of ketone (3-OHB) infusion; Dietary Supplement: Placebo - use of saline infusion

INTERVENTIONS:
Dietary Supplement: Hyperketonemia - use of ketone (3-OHB) infusion — The effect of intravenous ketone supplement
Dietary Supplement: Placebo - use of saline infusion — Saline is infused as an comparator

SUMMARY:
In the present study, patients with idiopathic pulmonary hypertension (IPAH) and chronic thromboembolic pulmonary hypertenion will be investigated in a randomized cross-over design with ketone infusions and placebo. Invasive and non-invasive hemodynamics will be evaluated

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a debilitating disease that affects both the pulmonary vasculature and the heart. It is associated with increased mortality and hospitalization and impairs daily life for the affected patients. Despite substantial advances in treatment within the past decade the prognosis remains poor with an 1-year mortality of more than 10%.1 The pathophysiology of PH is multifactorial and can be caused by left sided cardiac disease, pulmonary pathophysiological changes in the pulmonary vessels, respiratory diseases and pulmonary embolism.The treatment is targeted at the underlying cause. Hence, left sided heart disease is treated with anticongestive medications4 and respiratory disease by pulmonary medications. However, pulmonary vascular diseases such as chronic thromboembolic pulmonary hypertension (CTEPH) and idiopathic pulmonary arterial hypertension (IPAH) are treated with pulmonary endarterectomy and vasodilators targeting the pulmonary vasculature, respectively. However, not all patients have an optimal pulmonary hemodynamic response on treatment. If patients are left with persistent pulmonary hypertension the disease may progress further and cause right heart failure which worsens the prognosis.

Data from a recent study conducted at the investigator's institution demonstrated 40% increase in cardiac output during infusion of the ketone body 3-hydroxybutyrate (3-OHB). Intriguingly, this was associated with an increase in RV function and a decrease in the pulmonary vascular resistance of approximately 20%.

In the present study, 10 patients with IPAH and 10 patients with CETPH will be subjected to placebo and 3-OHB infusion in a randomized cross-over design. Each of the infusions will be given for 2.5 hours and cross-over will be carried out on the same day. Echocardiography and right sided heart catheterization will be applied and blood will be sampled.

ELIGIBILITY:
Inclusion Criteria:

* Persistent pulmonary hypertension (defined as PVR > 3 WU, pulmonary capillary wedge pressure (PCWP) < 15 mmHG, mean pulmonary arterial pressure (mPAP) ≥25 mmHg) on the most resent right heart catheterization.
* Preserved left ventricular ejection fraction (<50%) on most recent echocardiography
* Able to give informed consent

Exclusion Criteria:

* Other Significant pulmonary, mitral or aortic valve disease
* Other disease or treatment making subject unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Cardiac output (L/min | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Measured by Swan-Ganz monitoring

SECONDARY OUTCOMES:
mixed venous saturation (%) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Hemodynamics - Swan Ganz monitoring
systemic blood pressure (mmHg) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Hemodynamics - non-invasive blood pressure measurement
pulmonary capillary pressure (mmHg) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Hemodynamics - Swan Ganz monitoring
Pulmonary pressure (mmHg) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Hemodynamics - Swan Ganz monitoring
TAPSE (mm) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Echocardiography
RV strain (%) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Echocardiography
LV strain (%) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Echocardiography
systolic tricuspid plane velocity (cm/sec) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Echocardiography
Left ventricular ejection fraction (%) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Echocardiography
Changes in Prostaglandines (pmol/L) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Blood samples
pH | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Blood samples
sodium (mM) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Blood samples
potassium (mM) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Blood samples
lactate (mM) | changes during the infusion for 2.5 hours compared to 2.5 hours of Saline infusion
  Blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Roni R Nielsen, MD PhD, Principal Investigator — Dept. of Cardiology, Aarhus University Hospital
Locations (1):
- Dept. of cardiology, Aarhus University hospital Skejby,, Aarhus, Region Midjylland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen R, Christensen KH, Gopalasingam N, Berg-Hansen K, Seefeldt J, Homilius C, Boedtkjer E, Andersen MJ, Wiggers H, Moller N, Botker HE, Mellemkjaer S. Hemodynamic Effects of Ketone Bodies in Patients With Pulmonary Hypertension. J Am Heart Assoc. 2023 May 16;12(10):e028232. doi: 10.1161/JAHA.122.028232. Epub 2023 May 15. PMID 37183871